CLINICAL TRIAL: NCT06141642
Title: Self-Adaptive Immersive Virtual Reality Serious Game to Enhance Motor Skill Learning and Attention in Older Adults - A Double Blind Randomized Controlled Trial
Brief Title: Self-Adaptive Immersive Virtual Reality Serious Game to Enhance Motor Skill Learning and Attention in Older Adults
Acronym: SAVinGs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: #2020-1909
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Older Adults; Aging Well; Aging
Keywords: Aged

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-adaptive serious game (Experimental): Participants in this arm will follow, during three consecutive days, a serious game (REAsmashVR) intervention whose difficulty is automatically and progressively adapted to their motor and cognitive performance.
  REAsmashVR involves finding a target as fast as possible. The virtual target (a mole wearing a red miner's helmet) is presented with distractors (moles wearing different helmets). Participants use a controller to hit the target mole with a virtual hammer.
  In this arm, the REAsmashVR version uses a regulator to continuously moderate the location and timing of appearance of the target mole, the number and type of distractors and the working area. This regulator enables users to score 75% successful performance (driving motivation to play / learn).
  Interventions: Device: Self-adaptive serious game
- Non-adaptive serious game (Sham Comparator): Participants in this arm will follow, during three consecutive days, a serious game (REAsmashVR) intervention whose difficulty is not automatically adapted to their motor and cognitive performance.
  In this arm, the REAsmashVR version does not use a regulator to continuously adapt exercise difficulty according to user performance. Instead, the game randomly moderates the location of the target mole, the working area and the type of distractors. The appearance timing remains constant at 7 seconds, while the number of distractors gradually increases over time to simulate an adaptive game environment, ensuring participants are kept unaware of the intervention.
  Interventions: Device: Non-adaptive serious game

INTERVENTIONS:
Device: Self-adaptive serious game — A self-adaptive serious game in immersive virtual reality using the device MetaQuest 1 or 2
  Arms: Self-adaptive serious game
Device: Non-adaptive serious game — A non-adaptive serious game in immersive virtual reality using the device MetaQuest 1 or 2
  Arms: Non-adaptive serious game

SUMMARY:
While scientific evidence emphasizes the detrimental effect of sedentary behavior on health, the literature suggests that, on average, older adults spend 75% of their days in a sedentary manner, and often isolated (Petrusevski 2020). This lack of physical activity and social interaction not only leads to an increase in functional limitations and the risk of worsening an existing chronic disease but also elevates the risk of mortality. Furthermore, older adults face progressive functional decline, both in motor and cognitive aspects, as a result of aging, contributing to inactivity and sedentary behavior (Botö 2021).

The literature suggests that new technologies such as immersive virtual reality (iVR) and serious games serve as effective means to promote active leisure, thereby breaking isolation and reducing sedentary behavior. The development of these new technologies is also promising for objectively and quantitatively measuring motor and cognitive activity (e.g., kinematics, reaction time).

Serious games are defined as games whose primary objective is more focused on learning than entertainment. For instance, they allow the integration of physical and cognitive activity programs into a playful activity, conducive to long-term adherence. Their effectiveness is starting to be studied in hospitalized older adults (Cuevas-Lara 2021), especially as they also help combat age-related functional decline. Indeed, they provide the opportunity to promote and measure activity through enjoyable and self-administered exercises.

However, despite the growing interest in serious games, the impact of self-adaptive serious games, compared to traditional (non-adaptive) serious games, on motor skill learning and attention function in older adults remains unclear. This gap in knowledge necessitates a rigorous investigation. Therefore, this randomized controlled trial seeks to address this gap and achieve the following objectives:

1. Compare the effect of a self-adaptive serious game to a non-adaptive serious game on motor skill learning and attention in older adults.
2. Enhance the understanding of how motor skill learning in immersive virtual reality translates to older adults' activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Normal-to-corrected vision
* Score > 24 in the Montreal Cognitive Assessment
* Age > or = 65 years old

Exclusion Criteria:

* Severe comprehension issues
* History of seizures
* Prior experience with serious games in immersive virtual reality

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Motor function - Upper limb movement smoothness in immersive virtual reality | Day 1 (before intervention), day 2 and day 3 (at the end of the intervention)
  Spectral Arc Length (SPARC) of the normalized instant velocity signal
Motor function - Upper limb speed-accuracy trade-off in immersive virtual reality | Day 1 (before intervention), day 2 and day 3 (at the end of the intervention)
  This index is calculated by dividing the speed of performance by the accuracy of performance
Cognition - Response time in immersive virtual reality | Day 1 (before intervention) and day 3 (at the end of the intervention)
  Time between the target mole appearance and the and the successful hitting of the mole (in REAsmash VR evaluation module)
Cognition - Inhibition cost of response time in immersive virtual reality | Day 1 (before intervention) and day 3 (at the end of the intervention)
  Difference of response time between levels where the target mole is presented among non-salient distractors (levels 3 and 4), salient distractors (levels 1 and 2) and no-distractors (level 0) in REAsmashVR (evaluation module)

SECONDARY OUTCOMES:
Motor function - Coefficient of linearity in immersive virtual reality | Day 1 (before intervention), day 2 and day 3 (at the end of the intervention)
  Ratio between the ideal path (the length of the ideal route) and the distance covered by the controller
Motor function - Mean velocity in immersive virtual reality | Day 1 (before intervention), day 2 and day 3 (at the end of the intervention)
  Ratio between the distance covered by the controller and the duration of the task
Motor function - Peak velocity in immersive virtual reality | Day 1 (before intervention), day 2 and day 3 (at the end of the intervention)
  Highest instant velocity observed during the movement
Motor function - Coefficient of variation of the velocity in immersive virtual reality | Day 1 (before intervention), day 2 and day 3 (at the end of the intervention)
  Ratio between the standard deviation of the instant velocity and the mean velocity
Motor function - Lpath in immersive virtual reality | Day 1 (before intervention), day 2 and day 3 (at the end of the intervention)
  Total distance covered by the controller during the task
Motor function - Headpath in immersive virtual reality | Day 1 (before intervention), day 2 and day 3 (at the end of the intervention)
  Total distance covered by the headset during the task
Motor function transfer - Finger Nose Test | Day 1 (before intervention) and day 3 (at the end of the intervention)
  Motor-coordination test where participants are asked to touch their nose and a circular target (3 cm diameter) disposed on a wall 30cm away in the horizontal plane. Participants must realize as many repetitions as possible in 20s without missing the nose or the target.
Activity transfer - TEMPA_glass | Day 1 (before intervention) and day 3 (at the end of the intervention)
  The TEMPA (Test Évaluatif des Membres Supérieurs de Personnes Âgées) is an assessment designed to evaluate upper limb function in older adults, encompassing the performance of nine routine upper limb activities. Within the scope of this study, the investigators intend to assess participants' performance specifically in one of these tasks: pouring a glass of liquid and subsequently drinking it. The measurement will focus on the time taken by participants to complete this particular activity.
Activity transfer - Box and Block Test | Day 1 (before intervention) and day 3 (at the end of the intervention)
  The Box and Block Test (BBT) is a standardized performance-based assessment used to evaluate manual dexterity and upper extremity function, particularly in the context of gross motor skills. The test involves a wooden box divided into two compartments by a partition. Within one compartment, there are a certain number of wooden blocks. The objective of the test is to move as many blocks as possible from one side of the box to the other within 60s.
Cognition - Number of false positive in immersive virtual reality | Day 1 (before intervention) and day 3 (at the end of the intervention)
  The count of erroneously hit distractor moles in the VR evaluation module of REAsmash.
Cognition - Number of omissions in immersive virtual reality | Day 1 (before intervention) and day 3 (at the end of the intervention)
  The count of omitted target moles in the VR evaluation module of REAsmash.
Cognition transfer - Deary-Liewald reaction time task | Day 1 (before intervention) and day 3 (at the end of the intervention)
  A computerized test wherein participants are prompted to accurately respond to stimuli presented in either one or four squares at randomized intervals.

OTHER OUTCOMES:
Feasibility - Number of drop-outs | Day 1 (before intervention), day 2 and day 3 (at the end of the intervention)
  The count of participants that will not finish the experiment
Feasibility - Number of adverse events | Day 1 (before intervention), day 2 and day 3 (at the end of the intervention)
  The count of adverse events
Effectiveness of participants masking | Day 3 (at the end of the intervention)
  A Likert scale incorporating a confidence ratio, wherein participants are required to estimate and express their confidence level regarding the arm in which they were allocated
Participants' perception of immersive virtual reality and serious games | Day 3 (at the end of the intervention)
  Semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Charles Sebiyo Batcho, PT, PhD, Principal Investigator — Laval University
Locations (1):
- University Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Everard G, Vermette M, Dumas-Longpre E, Hoang T, Robitaille M, Sorrentino G, Edwards MG, Lejeune T, Batcho CS. Self-adaptive over progressive non-adaptive immersive virtual reality serious game to promote motor learning in older adults - A double blind randomized controlled trial. Neuroscience. 2025 Apr 6;571:7-18. doi: 10.1016/j.neuroscience.2025.02.053. Epub 2025 Feb 26. PMID 40021077